CLINICAL TRIAL: NCT00902005
Title: Endothelial Function, Inflammatory Disease Activity, and Bone and Cartilage Markers in RA and Spondyloarthritis Patients, Treated With TNFalpha-inhibitors in Combination With Methotrexate or Methotrexate or TNFalpha-inhibitors Alone - a Prospective Study
Brief Title: Endothelial Function, Inflammatory Disease Activity, and Bone and Cartilage Markers in Rheumatic Patients: The Influence of Antirheumatic Treatment
Acronym: PSARA
Status: Completed | Type: Observational
Sponsor: Revmatismesykehuset AS (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: S-07377b
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Ankylosing Spondylitis; Endothelial Dysfunction; Inflammatory Disease Activity
Keywords: Endothelial dysfunction; Bone and cartilage markers; Inflammatory disease activity; Rheumatoid arthritis; Psoriatic arthritis; Ankylosing Spondylitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Rheumatic patients: Three groups:
  RA patients: 30 starting on Methotrexate, 30 starting on combination of Methotrexate and TNFalpha inhibitor.
  PSA patients: 20 starting on Methotrexate, 20 starting on combination of Methotrexate and TNFalpha inhibitor.
  AS patients: 20 starting on TNFalpha inhibitor

SUMMARY:
The aim of this study is to examine the associations between inflammatory disease activity and endothelial function in rheumatoid arthritis (RA) and spondyloarthritis patients treated with methotrexate and Tumor Necrosis Factor alpha (TNFalpha)inhibitor in combination or methotrexate or TNFalpha-inhibitor alone. Further, to look for improvement in endothelial function, and decrease in bone and cartilage destruction during treatment with the combination therapy of TNFalpha-inhibitor and methotrexate in RA and Psoriatic Arthritis (PSA) patients. Last, examine the TNFalpha inhibitors influence on endothelial function and levels of bone and cartilage markers in patients with Ankylosing Spondylitis (AS).

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-80 years
* Able and willing to give written informed consent, and to comply with the requirements of the study protocol.
* Fulfilling the ACR 1987 revised diagnostic criteria for the diagnosis rheumatoid arthritis, or the diagnostic criteria by Moll and Wright for the diagnosis psoriatic arthritis, or the modified New York diagnostic criteria for ankylosing spondylitis.
* Clinical indication for starting treatment with methotrexate, TNFalpha- inhibitor or combination therapy.
* Use of reliable method of contraception for women with childbearing potential.

Exclusion Criteria:

* Lack of cooperativity
* Positive serology for hepatitis B or C
* History of positive HIV status.
* History of tuberculosis or untreated tuberculosis.
* PPD more than 15 mm in previously BCG immunized subjects. PPD 6 mm or more if not previously BCG immunized.
* Histoplasmosis or Listeriosis
* Persistent or recurrent infections
* Any inflammatory disease of permanence not related to RA, PSA or AS.
* Pregnancy or breast-feeding.
* Use of prednisolone more than 10 mg daily for 2 weeks at inclusion.
* Use of TNFalpha-inhibitor the last 4 weeks.
* History of cancer.
* Uncontrolled diabetes.
* Congestive heart failure (Nyha 3-4)
* Recent stroke (within 3 months)
* Previous diagnosis or signs of central nervous system demyelinating disease.
* Previously diagnosed immunodeficiency.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RA and spondyloarthritis starting with either combination therapy of TNFalpha-inhibitor and methotrexate or methotrexate or TNFalpha-inhibitor alone, at Lillehammer Hospital for Rheumatic diseases.Decision about treatment modality will be based on conventional clinial judgement.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2008-04; Primary Completion 2011-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To examine the association between inflammatory disease activity and endothelial function in RA and spondyloarthritis patients treated with methotrexate and TNFalpha-inhibitor in combination or methotrexate or TNFalpha-inhibitor alone | Baseline (before treatment starts), 6 weeks and 6 months after starting treatment

SECONDARY OUTCOMES:
CRP (C-reactive protein) | Baseline (before starting treatment), 6 weeks, 6 months after starting treatment
DAS28 (Disease activity score) | Baseline (before starting treatment), 6 weeks, 6 months after starting treatment
COMP (cartilage oligomeric matrix protein 1) | Baseline (before starting treatment), 6 weeks, 6 months after starting treatment
IL-6 (interleukin 6) | Baseline (before starting treatment), 6 weeks, 6 months after starting treatment
s-RAGE (Receptor of Advanced Glycation End products) | Baseline (before starting treatment), 6 weeks, 6 months after starting treatment

CONTACTS AND LOCATIONS:
Overall Officials: Knut Mikkelsen, MD, Study Chair — Lillehammer Hospital for Rheumatic Diseases; Gunnbjørg Hjeltnes, MD, Principal Investigator — Lillehammer Hospital for Rheumatic Diseases
Locations (1):
- Lillehammer Hospital for Rheumatic Diseases, Lillehammer, Oppland, Norway

REFERENCES:
- [Derived] Hokstad I, Deyab G, Wang Fagerland M, Lyberg T, Hjeltnes G, Forre O, Agewall S, Mollnes TE, Hollan I. Tumor necrosis factor inhibitors are associated with reduced complement activation in spondylarthropathies: An observational study. PLoS One. 2019 Jul 23;14(7):e0220079. doi: 10.1371/journal.pone.0220079. eCollection 2019. PMID 31335881
- [Derived] Deyab G, Hokstad I, Whist JE, Smastuen MC, Agewall S, Lyberg T, Ronda N, Mikkelsen K, Hjeltnes G, Hollan I. Methotrexate and anti-tumor necrosis factor treatment improves endothelial function in patients with inflammatory arthritis. Arthritis Res Ther. 2017 Oct 17;19(1):232. doi: 10.1186/s13075-017-1439-1. PMID 29041979
- [Derived] Ronda N, Greco D, Adorni MP, Zimetti F, Favari E, Hjeltnes G, Mikkelsen K, Borghi MO, Favalli EG, Gatti R, Hollan I, Meroni PL, Bernini F. Newly identified antiatherosclerotic activity of methotrexate and adalimumab: complementary effects on lipoprotein function and macrophage cholesterol metabolism. Arthritis Rheumatol. 2015 May;67(5):1155-64. doi: 10.1002/art.39039. PMID 25605003
- [Derived] Hjeltnes G, Hollan I, Forre O, Wiik A, Lyberg T, Mikkelsen K, Agewall S. Relations of serum COMP to cardiovascular risk factors and endothelial function in patients with rheumatoid arthritis treated with methotrexate and TNF-alpha inhibitors. J Rheumatol. 2012 Jul;39(7):1341-7. doi: 10.3899/jrheum.111401. Epub 2012 Jun 1. PMID 22660798